CLINICAL TRIAL: NCT03662243
Title: Treatment for Reading and Writing Deficits Following Acquired Brain Injury
Status: Completed | Type: Observational
Sponsor: Quality Living, Inc. (Other)
Responsible Party: Principal Investigator, Karen Hux, Director of Research, Quality Living, Inc.
Other Study IDs: Reading/writing treatment
Record Dates: First submitted 2018-09-03; First posted 2018-09-07 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: Acquired Brain Injury; Alexia; Agraphia
MeSH Terms: conditions — Brain Injuries; Dyslexia; Agraphia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Acquired brain injury participants: People with acquired alexia and/or agraphia secondary to brain injury who participate in the reading/writing intervention.
  Interventions: Behavioral: Multicomponent reading and writing treatment

INTERVENTIONS:
Behavioral: Multicomponent reading and writing treatment — Intervention procedures incorporated into the program include drilling on sight words to improve immediate recognition of common words; engaging in Multiple Oral Reading procedures to increase reading fluency; practicing oral spelling of sight words to improve spelling accuracy; generating written sentences to improve accurate spelling and use of written conventions (e.g., punctuation, capitalization); and summarizing and subsequently writing sentences about read material to establish strategies to enhance reading comprehension and promote written expression.

SUMMARY:
Many people with acquired brain injuries have deficits in reading decoding, reading comprehension, and written expression. Alexia is a phenomenon in which a person who previously could read has trouble doing so after having sustained a brain injury; likewise, agraphia is an acquired writing problem affecting one or more aspects of written communication. Alexia and agraphia sometimes co-occur with one another and/or with other language challenges, but they can also occur as isolated phenomena. Methods to treat alexia and agraphia often focus on single intervention techniques that address aspects of reading or writing in isolation-such as matching written and spoken letters or letter sounds, performing choral reading, tracing letters, etc. Existing research suggests that the effectiveness of these techniques is limited. However, when used in combination, such techniques may promote improved reading and written communication skills. As such, the purpose of this research is to determine the extent to which a multicomponent intervention program improves the reading and writing capabilities of people with acquired alexia and/or agraphia.

ELIGIBILITY:
Inclusion Criteria:

* Survivor of acquired brain injury
* Exhibits alexia and/or agraphia
* Past or current client of Quality Living, Inc., Omaha, Nebraska
* Fluent speaker of English

Exclusion Criteria:

* Vision impairment prohibiting reading of 24-point text
* Auditory comprehension problems precluding understanding of consent/assent information

Ages: 14 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: People enrolled in rehabilitation programs at Quality Living in Omaha, Nebraska, who are between the ages of 14 and 70 years and who experience alexia and/or agraphia secondary to acquired brain injury.
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2018-08-30 (Actual); Primary Completion 2020-09-15 (Actual); Study Completion 2020-09-15 (Actual)

PRIMARY OUTCOMES:
Change in score on Word Attack subtest of the Woodcock-Johnson III Test of Achievement. | Change from baseline at 8 weeks
  Subtest raw sores range from 0 to 32,with higher scores indicating better performance.
Change in score on Passage Comprehension subtest of the Woodcock-Johnson III Test of Achievement. | Change from baseline at 8 weeks
  Subtest raw scores range from 0 to 47, with higher scores indicating better performance.
Change in score on Word Reading subtest of the Wide Range Achievement Test 4. | Change from baseline at 8 weeks
  Subtest raw scores range from 0 to 70, with higher scores indicating better performance.
Change in score on Spelling subtest of the Wide Range Achievement Test 4. | Change from baseline at 8 weeks
  Subtest raw scores range from 0 to 57, with higher scores indicating better performance.
Change in score on Test of Silent Reading Speed and Efficiency. | Change from baseline at 8 weeks
  Raw scores range from 0 to 70, with higher scores indicating better performance.

SECONDARY OUTCOMES:
Sight word decoding accuracy | One time per week for 8 weeks
  Percent of correct decoding on 315 words included in Dolch pre-primer, primer, kindergarten, first grade, second grade, third grade, and nouns lists. Each word is scored as correct or incorrect, and a percent correct score is computed based on this scoring.
Oral reading rate of passages | As the first of five tasks of each session for 8 weeks (each session is 1 hour).
  Words per minute (wpm) during independent oral reading of passages. The criteria for progression to subsequent passages is a reading rate of 80wpm or better.
Decoding errors during oral reading of passages | As the first of five tasks of each session for 8 weeks (each session is 1 hour).
  Percent of uncorrected word decoding errors in a specified passage. The criterion for progression to subsequent passages is fewer than 5% uncorrected words production errors.
Oral spelling of words | As the second of five tasks of each session for 8 weeks (each session is 1 hour).
  Number of words spelled correctly on lists containing 15 words each. Introduction of a new word list will occur only after a participant correctly spells all words on the current list.

CONTACTS AND LOCATIONS:
Overall Officials: Karen Hux, Ph.D., Principal Investigator — Quality Living, Inc., Omaha, Nebraska
Locations (1):
- Quality Living, Inc., Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No